CLINICAL TRIAL: NCT06187688
Title: Measuring Pain Intensity in Cesarean Delivery Patients: a Comparison of 5 Scales
Brief Title: Measuring Pain Intensity in Cesarean Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Associate Professor, Prince of Songkla University
Other Study IDs: 66-355-8-1
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Patients to complete a questionnaire on measurement of pain intensity.

SUMMARY:
Pain intensity is commonly measured in research and clinical settings.

Primary objective:

To evaluate psychometric properties (validity, reliability, and utility) of 5 pain measurement tools: a verbal 11-point NRS, the FPS-R, a 6-point VDS, an 11-point NRS, and a 100 mm VAS in a sample of cesarean section patients.

Secondary objectives:

To evaluate whether the (new) word "very severe pain" is easier for patients to understand in comparison to the (old) word "worst pain imaginable.

To evaluate whether the (new) word "overall pain" is easier for patients to understand in comparison to the (old) word "average pain".

DETAILED DESCRIPTION:
1. Participants will be invited to participate in this study. If they agree to get involved, they will be provided a printed information sheet that describes the study purposes and procedures. A. The participants will not be disturbed if they are sleeping, caring for their baby or actively receiving a health care service.

   B. The research team will not ask ward nurses to provide the information sheet to the participants because nurses are already overwhelmed by their assigned jobs to provide nursing care to patients.
2. A "research staff person" will describe the purpose and procedures of the study, voluntariness of participation, potential benefits and harms, and rights to withdraw from the study, as also described on the information sheet.

   A. Research staff persons = anesthetic nurses B. The research team will not ask ward nurses to describe the purpose and procedures of the study to the participants because nurses are already overwhelmed by their assigned jobs to provide nursing care to patients.
3. Time will be provided for participants to ask any questions, and the research staff person will answer any questions asked.

   A. Unlimited time will be provided for the participants to respond to the study questions and complete the study measures. B. The participants can choose to participate on another day during their admission.
4. Any individual agreeing to participate will be asked to read and sign an informed consent form.
5. Participants will then be asked to provide demographic data and information about their pain (via interview/via a paper-and-pencil questionnaire developed for this purpose). The information gathered will include: age, education level and pain characteristics.
6. The participants will be instructed on how to use each assessment tool, and information about the measures will be repeated up to 3 times if requested by a participant.
7. The participants will be asked to rate their (1) current pain intensity, (2) maximum/worst pain intensity experienced during the past week, (3) average pain intensity experienced during the past week, and (4) minimum/least pain intensity experienced during the last week, using all five of the aforementioned scales.
8. Each type of scale will be presented on a separate page and in random order (using a Latin square design), so those participants are not able to easily refer to their previous responses when responding to each scale.
9. Hence, all participants will provide 20 ratings.
10. If any participant is unable to use a measure or answers incorrectly to any measurement tool, the administrator will not note any incorrect use while the participants are completing the measures, nor will they attempt to correct any errors made by participants in using the scales (other than to repeat the instructions up to 3 times, if requested by the participant).
11. After participants have provided the 20 ratings using the 5 pain measurement tools, they will be asked if they do or do not have a preference for any one type of scale. If they do have a preference, they will be asked to identify the scale that they prefer over the others.
12. Participants are asked to describe their pain characteristics using their own words.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Endorsing having post-cesarean section pain in the first 72 hrs following the operation
* Can speak and write in Thai, as determined by an ability to answer details about demographic information
* No motor deficits in the hands that would interfere with their ability to respond to a paper-and-pencil questionnaire

Exclusion Criteria:

* Age less than 18 years old
* Lack of fluency in Thai
* Neurological disorder or psychiatric illness that would interfere with participation or ability to provide informed consent
* Refusal to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who undergo cesarean delivery.
Sampling Method: Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the psychometric properties of the Verbal 11-point Numerical Rating Score (VNRS) in cesarean section patients. | January 2024 - December 2025
  To evaluate the psychometric properties of the 11-point Verbal Numerical Rating Score (VNRS) which 0 means "no pain" and 10 means "worst pain imaginable" in a sample of cesarean section patients.
To evaluate the psychometric properties of the Faces Pain Scale - Revised (FPS-R) in cesarean section patients. | January 2024 - December 2025
  To evaluate the psychometric properties of the Faces Pain Scale - Revised (FPS-R) which comprises with 6 faces ranging from the first neutral face as "no pain" and the sixth face as "the most severe pain" in a sample of cesarean section patients.
To evaluate the psychometric properties of the 6-point Verbal Descriptive Scale (VDS) in cesarean section patients. | January 2024 - December 2025
  To evaluate the psychometric properties of the 6-point Verbal Descriptive Scale (VDS) ranging from no pain, very mild pain, mild pain, moderate pain, severe pain and very severe pain in a sample of cesarean section patients.
To evaluate the psychometric properties of the 11-point Numerical Rating Scale (NRS) in cesarean section patients. | January 2024 - December 2025
  To evaluate the psychometric properties of the 11-point Numerical Rating Scale (NRS) where 0 means "no pain" and 10 means "worst imaginable pain" in a sample of cesarean section patients.
To evaluate the psychometric properties of the 100 mm Visual Analog Scale (VAS) in cesarean section patients. | January 2024 - December 2025
  To evaluate the psychometirc properties of the 100 mm Visual Analog Scale (VAS) where 0 mm (left end of the line) represents "no pain" and 100 mm (right end of the line) represents "worst pain imaginable" in a sample of cesarean section patients.
To directly compare the psychometric properties of 5 pain measurement tools (VNRS, FPS-R, VDS, NRS and VAS in a sample of cesarean section patients. | January 2024 - December 2025
  To directly compare the psychometric properties of 5 pain measurement tools in a sample of cesarean section patients:
  1. the VNRS
  2. the FPS-R
  3. the VDS
  4. the NRS
  5. the VAS

SECONDARY OUTCOMES:
To compare the easiness to respond between the newly proposed words and the previously used words, using percentage of correct response. | January 2024 - December 2025
  To compare the easiness to respond between the newly proposed word (very severe pain) and the previously used word (worst pain imaginable), using percentage of correct response.
To compare the easiness to respond between the newly proposed words and the previously used words, using percentage of correct response. | January 2024 - December 2025
  To compare the easiness to respond between the newly proposed word (overall pain) and the previously used word (average pain), using percentage of correct response.

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request.